CLINICAL TRIAL: NCT00268346
Title: A Phase II Trial of ZD1839 (IRESSA®) for Patients With Recurrent or Metastatic Cancer of the Esophagus or Gastroesophageal Junction
Brief Title: Gefitinib in Treating Patients With Recurrent or Metastatic Esophageal or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Adelstein, MD, Principal Investigator, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF5538; P30CA043703 (NIH); CCF-5538 (Other: Cleveland Clinic IRB); ZENECA-1839IL/0234
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; recurrent esophageal cancer; squamous cell carcinoma of the esophagus; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZD1839 (Experimental)
  Interventions: Drug: ZD1839

INTERVENTIONS:
Drug: ZD1839 — ZD1839 treatment will be taken once a day PO, every day about the same time
  Other Names: IRESSA®; Gefitinib

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well gefitinib works in treating patients with recurrent or metastatic esophageal or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Explore the activity of single agent gefitinib, in terms of response rate, in a patient population with recurrent or metastatic esophageal or gastroesophageal junction cancer.

Secondary

* Assess the toxicity of this drug in these patients.

OUTLINE: Patients are stratified according to prior treatment (yes vs no).

Patients receive oral gefitinib once daily for at least 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 76 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed squamous cell carcinoma, adenocarcinoma, or large-cell undifferentiated carcinoma of the esophagus or gastroesophageal junction

  * Patients must have disease that is either metastatic (i.e., M1b by the definitions of the American Joint Committee on Cancer 1997 staging system) or recurrent after definitive therapy, and must be considered incurable by conventional treatments
  * Patients with small cell, or mixed small cell/non-small-cell histology are ineligible
  * Patients with lymphoma or sarcoma are also ineligible
* Disease must be measurable in at least one dimension by physical exam, x-ray, CT scan or MRI, ultrasound, or endoscopy

  * Measurable disease can be a previously irradiated lesion if disease growth has been documented in the lesion since completion of radiation therapy
  * An elevation in carcinoembryonic antigen (CEA) is not sufficient to use by itself in response assessment

PATIENT CHARACTERISTICS:

* ECOG Performance Status 0-1
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase and AST < twice normal
* Bilirubin < twice normal
* Calcium normal
* No known severe hypersensitivity to study drug or any of its excipients
* No clinical evidence of any other uncontrolled malignancy except adequately treated basal or squamous cell skin cancer or in situ cervical cancer
* Pregnant or nursing women are ineligible
* Fertile patients must use effective contraception
* No evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* No evidence of clinically active interstitial lung disease

  * Patients with chronic stable radiographic changes who are asymptomatic need not be excluded

PRIOR CONCURRENT THERAPY:

* Patients may not have received more than one previous systemic treatment regimen

  * Systemic treatment may have been given as part of definitive (adjuvant, neoadjuvant, concurrent, or sequential) management or for metastatic or recurrent disease
  * Previously untreated patients are also eligible
* No previous treatment with study drug or any other epidermal growth factor receptor (EGFR) antagonists
* More than 30 days since prior treatment with a non-approved or investigational drug
* At least 4 weeks must have elapsed since any surgery, radiation therapy, or chemotherapy administration
* Recovered from previous oncologic or other major surgery
* No concurrent barbiturates (e.g., phenytoin), carbamazepine, rifampicin, phenobarbital or Hypericum perforatum (St. John's wort)
* No concurrent surgery, radiation therapy, hormonal therapy, or other chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-10; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from April 2003 to January 2010 from medical clinic
Groups:
- No Prior Chem Therapy: Patients receive oral gefitinib once daily for at least 8 weeks in the absence of disease progression or unacceptable toxicity.
- Prior Chemotherapy: Patients may not have received more than one previous systemic treatment regimen. Systemic treatment may have been given as part of definitive (adjuvant, neoadjuvant, concurrent, or sequential) management or for metastatic or recurrent disease. Patients receive oral gefitinib once daily for at least 8 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | No Prior Chem Therapy | Prior Chemotherapy
Started | 18 | 40
Started Treatment | 18 | 40
Completed | 18 | 37
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Prior Chem Therapy | Prior Chemotherapy | Total
Number analyzed (Participants) | 18 | 40 | 58
Age, Continuous [Median (Full Range); unit: years] | 66 [45 to 82] | 58 [33 to 73] | 60 [33 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 15 | 33 | 48

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Complete or Partial Response Rate of Single Agent ZD1839 in a Patient Population With Recurrent or Metastatic Cancer of the Esophagus or Gastroesophageal Junction, Using the RECIST 1.0 Criteria.
Description: The overall response is the number of patients with the best response recorded in measurable disease (target lesions) from start to disease progression.Complete response is the number of patients with the disappearance of all target lesions. Partial response is the number of patients with larger than or equal to 30% decrease in sum of the longest diameters from baseline. Progressive disease is larger than or equal to 20% increase in sum of the longest diameters over the smallest sum observed or appearance of new lesions. Stable disease is neither PR nor PD criteria met.
Time Frame: at 8 weeks after initiation of treatment
Population: All patients enrolled were analyzed
Measure: Number; unit: participants
Groups:
- No Prior Therapy; Prior Chemotherapy: All patients will receive oral ZD1839 250 mg daily. Pill counts will be conducted at every visit to monitor compliance. Treatment will be continued for a minimum of 8 weeks.
Arm/Group | No Prior Therapy | Prior Chemotherapy
Number analyzed (Participants) | 18 | 40
participants | 1 [0.1 to 27.3] | 3 [1.6 to 20.4]
Statistical Analysis 1: Comparison: No Prior Therapy vs Prior Chemotherapy; In patients with prior chemotherapy, >25% response indicates efficacy and <10% indicates lack of efficacy. In patients with no prior chemotherapy, >45% response indicates efficacy and <25% indicates lack of efficacy. Using a 5% significance level, the study was designed to have 80% power to test each hypothesis; Test type: Superiority or Other; p < 0.05, binomial test for a single proportion; percentage response = 6.9

ADVERSE EVENTS:
Time Frame: From study start to 30 days after final treatment
Arm/Group | No Prior Chem Therapy | Prior Chemotherapy
Serious Adverse Events (participants affected / at risk) | 4/18 | 4/40
Other Adverse Events (participants affected / at risk) | 13/18 | 33/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Prior Chem Therapy (N=18) | Prior Chemotherapy (N=40)
death (General disorders) | 0 (0) | 1 (1)
hospitalization (General disorders) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Prior Chem Therapy (N=18) | Prior Chemotherapy (N=40)
Anorexia (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 20
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 4
Fatigue (General disorders) | 0 | 2
Mucositis/Stomatitis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes